CLINICAL TRIAL: NCT07326501
Title: Attitudes and Perceptions of Corresponding Authors From Top International Medical Journals Regarding the Use of Artificial Intelligence in the Scientific Process
Acronym: AISurvey6 A+
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Chirplast02
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Artificial Intelligence; Biomedical Research; Scientific Publishing; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Authors Survey Group: This label identifies the single cohort of participants, consisting of corresponding authors invited to complete the anonymous online survey. No comparison or control groups are included.
  Interventions: Other: observational survey

INTERVENTIONS:
Other: observational survey — This is an observational, non-interventional study based on an anonymous online questionnaire. No intervention is administered to participants.

SUMMARY:
"Artificial intelligence (AI), including large language models and conversational tools, is increasingly being used in medical research. These tools may assist researchers at different stages of the scientific process, such as generating research ideas, reviewing the literature, analyzing data, writing manuscripts, and preparing articles for publication. While interest in AI is growing rapidly, there is still limited information on how these tools are actually perceived and used by leading medical researchers. This study aims to better understand the attitudes, perceptions, and self-reported uses of artificial intelligence among corresponding authors who have published in six major international medical journals. These authors play a key role in shaping scientific standards and editorial practices, and their views are essential to understanding how AI may influence the future of medical research. Participants are invited to complete an anonymous online questionnaire that asks about their familiarity with AI tools, how and when they use or plan to use them in the research process, the potential benefits they perceive, and the concerns or limitations they identify. The survey also explores participants' expectations regarding transparency, ethical guidance, and journal policies related to the use of artificial intelligence in scientific work.The study is observational and does not involve any medical intervention or collection of personal or health-related data. Participation is voluntary, and responses are fully anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Participants without any disease, condition, or related symptoms are permitted to participate. This study is a non-clinical, observational survey focusing on attitudes and practices related to artificial intelligence in scientific research, not on health conditions.

Exclusion Criteria:

* Authors who are not corresponding authors.
* Students, residents, interns, or trainees without corresponding author status.
* Individuals not involved in biomedical or medical research activities.
* Individuals who decline to participate or do not complete the online questionnaire.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of corresponding authors who have published scientific articles in leading international medical journals. Participants are identified through publicly available publication data from six major journals (The New England Journal of Medicine, The Lancet, JAMA, Nature, Science, and The BMJ) and are invited to participate via professional email addresses. The population includes adult researchers from diverse biomedical and medical disciplines, with no geographic restriction.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported attitudes regarding the use of artificial intelligence in the scientific research process | At the inclusion
  Participants report their attitudes and perceptions regarding the use of artificial intelligence in the scientific research process through multiple-choice and Likert-scale items. Responses are analyzed descriptively; higher scores indicate more favorable attitudes toward the use of artificial intelligence.
Perceptions regarding the use of artificial intelligence in the scientific research process | At the inclusion
  Participants report their attitudes and perceptions regarding the use of artificial intelligence in the scientific research process through multiple-choice and Likert-scale items. Responses are analyzed descriptively; higher scores indicate more favorable attitudes toward the use of artificial intelligence.

SECONDARY OUTCOMES:
Self-reported patterns of use, regarding artificial intelligence tools in scientific research and publishing | At the inclusion
  Anonymous online questionnaire developed for this study Responses are collected using multiple-choice questions and Likert-scale items. Higher scores reflect greater reported use of artificial intelligence and more positive evaluations of its benefits, while higher concern scores reflect greater perceived risks or limitations
Perceived benefits regarding artificial intelligence tools in scientific research and publishing | At the inclusion
  Anonymous online questionnaire developed for this study Responses are collected using multiple-choice questions and Likert-scale items. Higher scores reflect greater reported use of artificial intelligence and more positive evaluations of its benefits, while higher concern scores reflect greater perceived risks or limitations
Risk regarding artificial intelligence tools in scientific research and publishing | At the inclusion
  Anonymous online questionnaire developed for this study Responses are collected using multiple-choice questions and Likert-scale items. Higher scores reflect greater reported use of artificial intelligence and more positive evaluations of its benefits, while higher concern scores reflect greater perceived risks or limitations
Expectations regarding artificial intelligence tools in scientific research and publishing | At the inclusion
  Anonymous online questionnaire developed for this study Responses are collected using multiple-choice questions and Likert-scale items. Higher scores reflect greater reported use of artificial intelligence and more positive evaluations of its benefits, while higher concern scores reflect greater perceived risks or limitations

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Alpes Maritimes, France